CLINICAL TRIAL: NCT00866138
Title: Phase II Study of AB1010 in Patients With Relapse or Refractory Multiple Myeloma With t(4/14) Translocation Expressing or Not Expressing FGFR3
Brief Title: Masitinib in Relapse or Refractory Multiple Myeloma With t(4/14) Translocation Expressing or Not FGFR3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB04019
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; t(4/14); relapsing; refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — masitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): masitinib (AB1010)
  Interventions: Drug: masitinib (AB1010)

INTERVENTIONS:
Drug: masitinib (AB1010) — masitinib 9 mg/kg/day per os

SUMMARY:
This phase 2 study was designed to assess the safety and efficacy of masitinib (AB1010) in patients with relapsing/refractory t(4;14) Multiple Myeloma. Response and progression were assessed according to the Bladé revised IMWG criteria1 from lowest point.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed multiple myeloma with a t (4; 14) translocation by FISH and PCR, expressing or not expressing FGFR3 identified by FACS
* Patients with Multiple Myeloma progressing or relapsing after at least two prior therapies (including conventional chemotherapy and/or high dose therapy) or who get a reduction of M-protein less than 75% within 3 months after a high dose treatment (Melphalan 200mg/m2) or after the plateau obtained for 3 months duration following to a conventional chemotherapy
* Patient with rapidly progressive disease with cytopenia and / or renal failure have to be stabilized with chemotherapy (if possible 3 cycles of VTD ( Bortezomib/Thalidomide/dexamethasone) or high dose Melphalan regimen followed by a 4 weeks washout period before the inclusion in the study.
* Patients must have a clearly detectable and quantifiable monoclonal M- component value (>5 g/l) in the serum and / or urine light chain excretion (>0,5 g/d)

Exclusion Criteria:

* Prior corticosteroids within two weeks before enrolment
* Prior local irradiation within two weeks before enrolment
* Prior experimental or standard treatment (other than steroids and local irradiation) within 30 days before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-02 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Tumor Response Rate, based on the criteria published by Blade and on the criteria SWOG | 16 weeks

SECONDARY OUTCOMES:
Tumor response rate with AB1010 plus dexamethasone | 16 weeks
Time to tumor progression and duration of response in responder patients | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Louis, Paris, France